CLINICAL TRIAL: NCT00906802
Title: Benefit of R-Y Reconstruction After Pancreaticoduodenectomy
Brief Title: Benefit of Roux-en-Y (R-Y) Reconstruction After Pancreaticoduodenectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kochi University (Other)
Responsible Party: Kochi Medical School, Kochi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RPD Study
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2009-07-23 (Estimated); Status verified 2009-07

CONDITIONS: Pancreatic Cancer
Keywords: pancreaticoduodenectomy; reconstruction
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- R-Y reconstruction (Experimental): the reconstruction was performed by R-Y anastomosis
  Interventions: Procedure: R-Y reconstruction
- conventional reconstruction (No Intervention): the anastomosis was performed by B-II

INTERVENTIONS:
Procedure: R-Y reconstruction — The reconstruction was performed by R-Y anastomosis.
  Other Names: the cutting R-Y anastmosis
  Arms: R-Y reconstruction

SUMMARY:
One of the most common complications of pancreaticoduodenectomy (PD) is delayed gastric emptying (DGE), otherwise known as "gastroparesis," which is not fatal but results in prolonged hospital stay and increased hospital costs. Delayed gastric emptying is defined as nasogastric decompression after postoperative day (POD) 10 or a failure to tolerate a regular diet after POD 14. The incidence of DGE has been reported to range from 5% to 72%.

DETAILED DESCRIPTION:
We hypothesized that the hand-sewn, two-layered, or continuous suture, could induce anastomotic edema to indeed the afferent peristalsis, which is one of the causes of DGE.

ELIGIBILITY:
Inclusion Criteria:

* These patients were to undergo elective pancreatic head resection for the treatment of periampullary mass

Exclusion Criteria:

* A body weight loss greater than 10% during the six months prior to surgery
* The presence of distant metastases
* Seriously impaired function of vital organs due to respiratory, renal or heart disease

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2003-04; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
the incidence of DGE | 3-6 months

SECONDARY OUTCOMES:
the incidence of other complication associated with reconstruction | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kazuhiro Hanazaki, Prof, Study Chair — Kochi University
Locations (1):
- Kochi Medical School, Nankoku, Kochi, Japan